CLINICAL TRIAL: NCT02786433
Title: Virtual Reality Effects on Functional Capacity and Quality of Life of People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Douglas Monteiro da Silva, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 18732713.0.0000.5193
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

ARMS (2):
- GROUP CONTROL (Active Comparator): Participants in the control group only underwent conventional physiotherapy. Conventional therapy includes stretching and strengthening exercises with cane aid, leggings , elastic band and overball for upper and lower limbs , in addition to gait and balance training.
  The intervention for the control group was applied for five weeks with sessions of 60 minutes twice a week
  Interventions: Other: conventional physiotherapy
- EXPERIMENTAL GROUP (Experimental): The subjects in the experimental group underwent conventional physiotherapy (The same applied in the control group) associated with virtual reality , performed with the console X -Box Kinect® of Microsoft. Durante the achievement of the virtual reality practice, Kinect and Kinect games Adventures® Dance® demanded the anterior movements players -posterior and lateral , as well as jumps and squats to get rid of the game obstacles. They Kinect Dance® game were all required movements of the previous game more dance . The intervention lasted five weeks , with two weekly sessions lasting 30 minutes to conventional therapy and 30 minutes to virtual reality.
  Interventions: Other: Virtual Reality with X- Box Kinect®

INTERVENTIONS:
Other: conventional physiotherapy
  Arms: GROUP CONTROL
Other: Virtual Reality with X- Box Kinect®
  Arms: EXPERIMENTAL GROUP

SUMMARY:
Introduction: Parkinson's disease (PD) is a progressive neurodegenerative disorder of dopaminergic neurons that can cause some mobility limitations and it has association with quality of life (QOL) in patients with PD. Virtual reality (VR) has been used to treat of these patients Objective: Evaluate the functional capacity and QOL of individuals with PD using VR with X-Box Kinect®. Methods: Were selected 20 individuals classified as stages 1-3, aged 50-75 years. They were divided by lot into two groups (control and experimental) with ten patients in each. The group (CG) treated with exercises (conventional therapy) during five-week, with two sessions per week lasting 60 minutes, while the experimental group (EG) spent half the time with conventional physical therapy and other half of time in virtual rehabilitation (VR). Subjects were evaluated before and after treatment using the following scales: Unified Parkinson's Disease Rating Scale and Parkinson's Disease Questionnaire .

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of idiopathic Parkinson's disease
* Male and female
* Stage 1-3 of the Hoehn and Yahr scale.

Exclusion Criteria:

* Have other neurological diseases
* They have decompensated systemic diseases
* Musculoskeletal changes that prevent the achievement of movements
* With lowering of the cognitive level assessed using the MiniMental State examination with cutoff point according to education
* With respiratory impairment
* With medical restrictions for performing exercises
* In physical therapy, occupational therapy service for 3 months or more;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale - Evaluates disease progression | 8 weeks
  Through the UPDRS disease progression was evaluated. Composed of 42 items, divided into four parts: mental activity, behavior and mood ; activities of daily living, motor operation and complications of drug therapy. For this study we evaluated the items : activities of daily living and motor examination on . The score for each item ranges from 0 to 4, and the maximum value indicates greater involvement by the disease and the minimum normality.
Parkinson's Disease Questionnaire (PDQ-39) - evaluates quality of life | 8 weeks
  The PDQ-39 is a method that evaluates the quality of life (QOL) in patients with PD through a questionnaire self-explanatory and easy to understand. There are 39 items divided into eight categories: mobility; activities of daily living; emotional well-being; social difficulties of PD; social support; cognition; communication and bodily discomfort. The score ranges from 0 (no problem) to 100 (maximum problem), or a low score indicates a better perception of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Pernambuco Parkinson Association, Recife, Pernambuco, Brazil